CLINICAL TRIAL: NCT03859128
Title: A Phase II/III, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Toripalimab (Recombinant Humanized Anti-PD-1 Monoclonal Antibody, JS001) Versus Placebo as Adjuvant Therapy in Patients With Hepatocellular Carcinoma at High Risk of Recurrence Following Radical Resection
Brief Title: Toripalimab or Placebo as Adjuvant Therapy in Hepatocellular Carcinoma After Radical Resection
Acronym: JUPITER 04
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-016-III-HCC
Record Dates: First submitted 2019-02-18; First posted 2019-03-01 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): TORIPALIMAB 240mg ,Q3W, up to 16 cycles
  Interventions: Biological: TORIPALIMAB INJECTION(JS001 )
- Group B (Placebo Comparator): Placebo 240mg Q3W, up to 16 cycles
  Interventions: Biological: TORIPALIMAB INJECTION(JS001 )

INTERVENTIONS:
Biological: TORIPALIMAB INJECTION(JS001 ) — Arm A: Toripalimab 240mg IV(Injection of Vein) Q3W Arm B: Placebo 240mg IV(Injection of Vein) Q3W

SUMMARY:
This study will investigate if Toripalimab (A PD-1 Inhibitor) will improve recurrence-free survival (RFS) compared to placebo in participants with HCC and are at high risk of recurrence after complete resection with no residual of tumour.

ELIGIBILITY:
Inclusion Criteria:

1. HCC with at least one protocol defined risk factor, diagnosed confirmed by central pathological review and received R0 resection;
2. BICR confirmed no resdual tumor lesions are detected in liver;
3. Child-Puch score, Class A;
4. ECOG score is 0;

Exclusion Criteria:

1. Patients previously received PD-1 antibody, PD-L1 antibody, PD-L2 antibody or CTLA-4 antibodies, including those who have participated in the JS001 clinical study;
2. Portal vein tumor thrombi or liver metastases or recurrent liver cancer;
3. With symptoms of central nervous system metastasis;
4. With any history of active autoimmune disease or autoimmune disease;
5. Known liver diseases with clinical significance;
6. Patients infected by hepatitis B virus (HBV), hepatitis C virus (HCV), hepatitis D virus (HDV):

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-04-18 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
BICR-RFS | Time frame is up to 31 months (for interim analysis, up to 44 months for Primary analysis)
  Defined as the time from randomization to the first documented disease recurrence or death.

SECONDARY OUTCOMES:
Investigator-RFS | up to 44 months
  the time from randomization to the date of the first documented progressive disease (tumor evlauation by BICR in accordance with RECIST 1.1), or to the date of death for any cause, whichever occurs first
12-month recurrence-free survival rate (RFS12) | up to 44 months
  probability of patients without recurrence or death for any cause at Month 12
24-month recurrence-free survival rate (RFS24) | up to 44 months
  probability of patients without recurrence or death for any cause at Month 24
Time to recurrence (TTR) | up to 44 months
  the time from randomization to the first documented disease recurrence
Time to local recurrence (TTLR) | up to 44 months
  the time from randomization to the first documented local disease recurrence
Overall survival (OS) | up to 44 months
  the time from randomization to death for any cause
12- and 24-month overall survival rate (OS12 and OS24) | up to 44 months
  probability of patients surviving at Month 12 and 24, respectively
Incidence of AEs | up to 44 months
  Incidence of AEs (including SAEs and AESIs) is evaluated by the investigator, and severity is determined in accordance with CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality, China